CLINICAL TRIAL: NCT07191743
Title: Assessment of Physical Function in Critically Ill Patients With the Chelsea Critical Care Assessment Tool (CPAX)
Brief Title: Functional Assessment in Critically Ill Patients
Status: Recruiting | Type: Observational
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Hospital Universitario Pedro Ernesto (Other); Instituto Nacional de Infectologia Evandro Chagas (Unknown)
Responsible Party: Principal Investigator, Jose Roberto Lapa e Silva, Full Professor of Pneumology, Universidade Federal do Rio de Janeiro
Other Study IDs: 65516422.7.0000.5259
Record Dates: First submitted 2025-08-26; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Intensive Care Unit Acquired Weakness; Intensive Care Unit (ICU) Acquired Weakness (ICU - AW)
Keywords: Critical Care; Intensive Care Units; Physical Therapy Department, Hospital; Muscle Weakness; Functional Status; Physical Functional Performance; Outcome Assessment, Health Care; Rehabilitation
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survivors: Adult patients admitted to the general ICU at Pedro Ernesto University Hospital (HUPE) who were discharged from the ICU to the hospital ward.
- Non-Survivors: Adult patients admitted to the general ICU at Pedro Ernesto University Hospital (HUPE) who died during their ICU stay.

SUMMARY:
This longitudinal, prospective observational study aims to evaluate functional status in critically ill adult patients in the Intensive Care Unit using the Chelsea Critical Care Physical Assessment Tool (CPAx). The primary objective is to analyze CPAx score variation as a potential predictor of clinical outcomes, including mortality and duration of mechanical ventilation. Functional assessments will be performed at intensive care unit (ICU) admission and discharge to monitor changes in physical function and to predict adverse clinical outcomes.

DETAILED DESCRIPTION:
This prospective, longitudinal, and observational study will be conducted at the general ICU of Pedro Ernesto University Hospital (HUPE). Demographic and clinical information at admission will be collected, including age, sex, type of airway at ICU admission, cause of ICU admission, comorbidities, and clinical scores such as Sepsis-related Organ Failure Assessment (SOFA), Simplified Acute Physiology Score III (SAPS III), and Charlson Comorbidity Index. During the ICU stay, data on the use of invasive mechanical ventilation, non-invasive ventilation, high-flow nasal cannula (HFNC), renal replacement therapy, extubation, and reintubation will be recorded. The CPAx will be assessed at ICU admission and discharge. Additionally, total hospital and ICU length of stay, as well as days on mechanical ventilation, will be recorded.The study aims to analyze the variation in CPAx scores as a predictor of adverse clinical outcomes, including mortality and duration of mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria: All adult patients admitted to the Pedro Ernesto University Hospital (HUPE) General ICU over 18 years of age and with an ICU stay greater than or equal to 48 hours will be included.

Exclusion Criteria:

* Pregnancy
* Inability to record the CPAx score within the first 48 hours of ICU admission or on the day of ICU discharge
* ICU readmission
* Known comorbidities causing generalized weakness, such as neuromuscular or neurological diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The general ICU admits both surgical patients and clinical patients, including those with acute illnesses or decompensations of chronic diseases. Participants include both male and female patients.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
hospital mortality | 12 months
  Mortality will be collected during the period of hospitalization

SECONDARY OUTCOMES:
mechanical ventilation days | 6 months
  It will be collected from the date of intubation in the intensive care unit until the date of extubation or up to 48 hours off mechanical ventilation in cases of tracheostomized patients and/or until the outcome of death
ICU length of stay | 6 months
  It will be collected from the date of intensive care unit admission until the outcome of discharge from the intensive care unit or death.
length of hospital | 12 months
  It will be collected from the date of intensive care unit admission until the outcome of hospital discharge or death.
Extubation rate | 30 days
  Proportion of patients who were extubated during ICU stay.
Reintubation rate | 30 days
  Proportion of patients who require reintubation after extubation during ICU stay.

CONTACTS AND LOCATIONS:
Overall Officials: PEDRO L SILVA, PhD, Study Director — Pulmonary Investigation Laboratory, Carlos Chagas Filho Institute of Biophysics (IBCCF), Federal University of Rio de Janeiro (UFRJ)
Locations (1):
- Pedro Ernesto University Hospital, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No